CLINICAL TRIAL: NCT06752564
Title: Effects of a Goal-Oriented Care Interventions on Self-efficacy, Symptom Disorder, and Quality of Life in Patients with Multiple Chronic Diseases
Brief Title: Impact of Goal-Directed Care Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202301193B0
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Multiple Chronic Diseases
Keywords: quality of life; symptom disorder
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): The experimental group during hospitalization additionally received 40 minutes of one-on-one education three times a week for three weeks, as the Goal-Oriented Care program for 6 hours in total, followed by telephone sessions of 20 minutes every month for six months post-discharge.
  Interventions:
  Behavioral: The Goal-Oriented Care program Behavioral: The routine health education
  Interventions: Behavioral: Goal-Oriented Care Model; Behavioral: standard health education
- The control group : standard health education (Active Comparator): The control group received standard health education. The content of the standard health education included verbal instructions provided by nurses during the general hospital stay, as well as the distribution of educational pamphlets. These instructions covered topics such as the frequency of dialysis and dietary control. The standard health education was generic, without a specific schedule or structured content.
  Interventions: Behavioral: standard health education

INTERVENTIONS:
Behavioral: Goal-Oriented Care Model — The experimental group : Goal-Oriented Care (GOC) The concept of Goal-Oriented Care (GOC) was first introduced by Mold et al. in 1991, addressing the limitations of problem-oriented care, which focuses on eradicating diseases and preventing death. GOC is defined as a process of reaching a consensus on health-related goals between the healthcare team and the patient (Vermunt et al., 2017). It is based on patients' core values and priorities within a clinical context, guiding medical interventions and specific treatment decisions (Secunda et al., 2020).
  Healthcare professionals using GOC aim to help patients achieve their maximum personal health potential, aligning care with individual goals. The clear direction provided by GOC fosters teamwork and interdisciplinary collaboration (Gray et al., 2020). When establishing long-term goals with patients, it is crucial to revisit and adjust these goals, considering realistic survival timelines, as time plays a vital role in goal-setting.
  Arms: Experimental
Behavioral: standard health education — The control group received standard health education. The content of the standard health education included verbal instructions provided by nurses during the general hospital stay, as well as the distribution of educational pamphlets. These instructions covered topics such as the frequency of dialysis and dietary control. The standard health education was generic, without a specific schedule or structured content.

SUMMARY:
Abstract The study explores the effects of a goal-directed care intervention on self-efficacy, symptom distress, and quality of life in patients with multiple chronic conditions.

Objective:

To evaluate whether patients with multiple chronic conditions exhibit significant improvement in self-efficacy after receiving a goal-directed care intervention compared to their pre-intervention status.

To assess whether symptom distress is significantly reduced following the intervention.

To determine whether patients experience a significant enhancement in quality of life post-intervention.

Background:

Global population aging is an ongoing phenomenon with increasing impact worldwide. According to the United Nations Population Report, the average global age in 2019 was 28 years and is projected to rise by 10 years to 38 years by 2050. The proportion of the population aged 65 and above grew from 8% in 1950 to 11% in 2009, and it is expected to reach 22% by 2050.

With advances in healthcare quality, the challenges of an aging population are intensifying. Problem-oriented care models, while widely used, are time-intensive and contribute to increased complexity in clinical practice. In contrast, a goal-directed care model focuses on patient-centered outcomes that align with individual priorities rather than addressing each disease separately. This approach reduces conflict and workload for clinical teams while enhancing trust and satisfaction among patients.

Goal-directed care is particularly beneficial for patients with multiple chronic conditions, who often face conflicting care options. This study highlights the potential of such an approach to streamline care delivery and improve outcomes in self-efficacy, symptom management, and overall quality of life.

DETAILED DESCRIPTION:
1. Multiple Chronic Conditions (MCC) Multiple Chronic Conditions (MCC), also known as multimorbidity, is defined as the co-occurrence of two or more chronic diseases, affecting 55% to 98% of the U.S. population aged 65 and older. The terms "multiple chronic conditions" and "multimorbidity" are often used interchangeably. Although MCC is a relatively recent concept, it has been recognized as a MeSH term since 2015. The prevalence of MCC is increasing, especially among the elderly. Studies show that 32% of patients in general practice in the Netherlands have MCC, and approximately 40-60% of older adults across Europe experience MCC.

   The high prevalence and management challenges of MCC in the context of an aging population signal an impending public health crisis. Older adults with MCC are more susceptible to adverse effects from conditions such as hypertension, cardiovascular disease, diabetes, and dementia. In the United States, healthcare costs for individuals aged 65 and older are three times higher than for working-age adults and five times higher than for children. Managing chronic diseases significantly increases healthcare costs, even in advanced healthcare systems, with the annual expenses for diagnosis and treatment continuing to rise .
2. Goal-Oriented Care (GOC) The concept of Goal-Oriented Care (GOC) was first introduced by Mold et al. in 1991, addressing the limitations of problem-oriented care, which focuses on eradicating diseases and preventing death. GOC is defined as a process of reaching a consensus on health-related goals between the healthcare team and the patient . It is based on patients' core values and priorities within a clinical context, guiding medical interventions and specific treatment decisions.

   Healthcare professionals using GOC aim to help patients achieve their maximum personal health potential, aligning care with individual goals. The clear direction provided by GOC fosters teamwork and interdisciplinary collaboration. When establishing long-term goals with patients, it is crucial to revisit and adjust these goals, considering realistic survival timelines, as time plays a vital role in goal-setting.

   GOC is especially relevant for managing patients with high disease complexity, offering benefits such as:

   Promoting patient autonomy and person-centered care. Avoiding unnecessary care processes and identifying valuable care components. Providing psychological care for patients and emotional support for their families.
3. Self-Efficacy Self-efficacy refers to an individual's confidence in their ability to perform behaviors that lead to desired outcomes. It is a mechanism for effective self-management, particularly for elderly individuals with chronic diseases, helping to reduce complications, injuries, and premature death while enabling normal social functioning.

   Measuring self-efficacy provides a standardized and convenient method for assessing patients' self-management potential, recommended as part of chronic disease care management. Patients with MCC often face challenges in self-management due to conflicting care plans from various providers. Enhancing self-efficacy through self-management support is associated with improved outcomes, including better quality of life.
4. Symptom Distress Patients with MCC frequently experience difficulty managing their symptoms, making symptom self-assessment crucial for health management. The persistence and severity of symptoms are significant determinants of healthcare utilization. However, symptoms can be challenging to interpret, and physicians may focus solely on symptom relief, sometimes overlooking the patient's broader symptom experience.

   Symptom management aims to reduce frequency and severity while alleviating distress through biomedical, professional, and management strategies . In Taiwan, the prevalence of physical symptom distress is 5%, with women more affected than men. Symptom distress is associated with higher rates of anxiety, depression, and healthcare utilization.
5. Quality of Life (QoL) Health-related quality of life (HRQoL) focuses on the impact of diseases, injuries, or treatments on physical function and their subsequent effects on physical, psychological, and social dimensions. QoL is inherently subjective and can be defined by individual satisfaction with economic status, health, and life conditions.

For elderly individuals, managing chronic diseases significantly affects QoL by increasing care pressures and reducing independence. Studies indicate that higher education levels and better financial status positively influence QoL by enhancing self-esteem and empowerment.

Research Methods This study adopts an experimental design conducted in a 3D integrated medical ward. Participants are hospitalized patients with MCC, referred by physicians or specialist nurses based on inclusion criteria. Eligible patients are randomly assigned to a control or experimental group.

The control group receives standard health education, including verbal instructions and printed materials on diet and treatment frequency. The experimental group receives additional "Goal-Oriented Care" intervention courses, focusing on self-efficacy, symptom distress, and QoL. Structured questionnaires are used pre- and post-intervention to evaluate the program's effectiveness.

Intervention Measures The GOC intervention centers on patient-focused goals, incorporating patients' and families' priorities. Using motivational interviewing, the healthcare team educates patients on disease management and the importance of self-efficacy, symptom management, and QoL. Education materials include booklets and visual aids to facilitate understanding. The intervention fosters trust and collaboration among patients, families, and the healthcare team to improve outcomes in MCC management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with two or more chronic diseases.
* Age ≥ 20 years and < 80 years.
* Clear consciousness and ability to communicate in Mandarin or Taiwanese dialect.
* Patients who consent to participate in the study after being informed of its purpose.

Exclusion Criteria:

* Presence of mental health disorders such as schizophrenia
* Bipolar disorder
* Major depressive disorder, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health Self-Efficacy | After the patient signs the informed consent form, basic demographic data, laboratory reports, and structured questionnaires (self-efficacy, symptom distress, and quality of life) will first be collected. Before intervention program.
  The measure of self-efficacy evaluates patients with multiple chronic illnesses, reflecting their confidence in performing specific health-related activities. Participants respond to statements such as, "I am confident that I can eat regularly," or "I can exercise without the company of others." Scores for these health management-related items range from 1 (no confidence at all) to 100 (completely confident).
Symptom Distress Scale | After the patient signs the informed consent form, basic demographic data, laboratory reports, and structured questionnaires (self-efficacy, symptom distress, and quality of life) will first be collected. Before intervention program.
  The "Symptom Distress Scale," developed by Lai (1998), is used to assess the severity of symptom distress perceived by the patient.
  The scale, collaboratively designed by the original author and three experienced cancer clinical care professionals, includes 22 common symptoms faced by cancer patients: nausea, vomiting, appetite issues, insomnia, pain, fatigue, bowel movements, urination, shortness of breath, coughing, bloating, dry mouth, oral/esophageal pain and ulceration, anxiety, concentration problems, appearance, bleeding, shivering/temperature fluctuations, fever, numbness, chest tightness, and heartburn.
  The scale uses a five-point Likert scoring system:
  1. point: "No distress"
  2. points: "Mild distress"
  3. points: "Moderate distress"
  4. points: "Severe distress"
  5. points: "Very severe distress" Scores range from 22 to 110, with higher scores indicating greater levels of symptom distress. In this study, the Cronbach's alpha coefficient for the sample was 0.78.
  The Taiwanese Somat
Quality of Life Scale | After the patient signs the informed consent form, basic demographic data, laboratory reports, and structured questionnaires (self-efficacy, symptom distress, and quality of life) will first be collected. Before intervention program.
  The Taiwanese version of the Short Form-36 (SF-36) is a self-reported tool that evaluates health-related quality of life (QoL) across eight dimensions:
  Physical Functioning (PF) Role Limitations Due to Physical Health (MR) Bodily Pain (BP) General Health (GH) Vitality (V) Social Functioning (SF) Role Limitations Due to Emotional Problems (EP) Mental Health (MH)
  Each dimension is scored from 0 to 100, where 100 represents excellent health and 0 indicates poor health. The SF-36 includes 36 items corresponding to 8 health domains, divided into two main components:
  Physical Component Summary (PCS), which includes physical functioning, role limitations due to physical health, bodily pain, and general health.
  Mental Component Summary (MCS), which includes vitality, social functioning, emotional role, and mental health.
  Scores range from 0 to 100, with 0 indicating extremely poor health and 100 indicating perfect health.

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No